CLINICAL TRIAL: NCT07396168
Title: Nemolizumab to Treat Lichen Planopilaris, a Noncontrolled, Prospective, Pilot Study.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Skin Center Dermatology Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NemoLPP
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lichen Plano-Pilaris
MeSH Terms: conditions — Lichen Planus | interventions — nemolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receive nemolizumab injections every 4 weeks, weight based dosing (Experimental)
  Interventions: Drug: Nemolizumab

INTERVENTIONS:
Drug: Nemolizumab — subcutaneous injection

SUMMARY:
Lichen planopilaris (LPP) is a primary lymphocytic cicatricial alopecia characterized by progressive, permanent hair loss and scalp symptoms such as pruritus and burning. Current treatments-including topical and intralesional corticosteroids, hydroxychloroquine, and immunosuppressants-are often inadequate, with limited evidence for efficacy and frequent treatment switching or discontinuation due to side effects or lack of response.1,2 Recent systematic reviews and meta-analyses highlight the need for new, targeted therapies. 3,4 Nemolizumab, an IL-31 receptor antagonist, FDA-approved for prurigo nodularis and atopic dermatitis, has demonstrated efficacy in pruritic and fibrosing dermatoses, making it a rational candidate for LPP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Clinical and/or histopathologic diagnosis of LPP.
* Presence of scalp pruritus.
* Average Peak Pruritus Numerical Rating Scale (PP-NRS) score ≥4 in the 7 days prior to Day 1.
* Ability and willingness to provide written informed consent and comply with study procedures.
* Willingness to undergo optional scalp biopsy for research purposes.

Exclusion Criteria:

* Other forms of alopecia that may interfere with study assessments.
* Any systemic disease associated with hair loss.
* Inflammatory or infectious scalp disease that may interfere with the study.
* Any other conditions associated with pruritus.
* Prior use of nemolizumab.
* Current treatment with systemic or topical JAK inhibitors or biologics (unless appropriate washout period completed; minimum 12 weeks).
* Current treatment with DMARDs (unless appropriate washout period completed; minimum 12 weeks).
* Prior treatment failure of scarring alopecia with systemic or topical JAK inhibitors or
* biologics.
* Current treatment with topical or intralesional corticosteroids (unless appropriate washout period completed; minimum 4 weeks).
* Any other current treatments for hair loss (e.g., oral/topical minoxidil, PRP) unless stable for at least 6 months or 3 months washout completed.
* Allergy or hypersensitivity to nemolizumab or any excipients.
* Pregnancy or unwillingness to use highly effective contraception.
* Any medical condition that, in the opinion of the investigator, may interfere with study participation or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at 24 weeks in Lichen Planopilaris Activity Index (LPPAI) | 24 weeks
Change from baseline at 24 weeks in Investigator Global Assessment (IGA) score (scarring alopecia version) | 24 weeks

SECONDARY OUTCOMES:
Change from baseline at 24 weeks in Peak Pruritus NRS. | 24 weeks

OTHER OUTCOMES:
Change from baseline at 24 weeks in hair count and average hair shaft thickness (digital trichoscopy). | 24 weeks
Incidence and severity of treatment-emergent adverse events. | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Skin Center Dermatology Group, New City, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmadi Kahjoogh H, Yazdanian N, Behrangi E, Roohaninasab M, Hejazi P, Goodarzi A. Efficacy, safety, tolerability, and satisfaction of N-acetylcysteine and pentoxifylline in lichen planopilaris patients under treatment with topical clobetasol: A triple arm blinded randomized controlled trial. Dermatol Ther. 2022;35(8). doi:10.1111/dth.15639
- [Background] Cho BK, Sah D, Chwalek J, et al. Efficacy and safety of mycophenolate mofetil for lichen planopilaris. J Am Acad Dermatol. 2010;62(3):393-397. doi:10.1016/j.jaad.2009.05.018
- [Background] Fatemi Naeini F, Mohaghegh F, Jelvan M, Asilian A, Saber M. Cyclosporine or methotrexate, which one is more promising in the treatment of lichen planopilaris?; A comparative clinical trial. Int Immunopharmacol. 2020;86:106765. doi:10.1016/j.intimp.2020.106765
- [Background] Lajevardi V, Ghiasi M, Balighi K, et al. Efficacy and safety of oral pioglitazone in the management of lichen planopilaris in comparison with clobetasol: A randomized clinical trial. Dermatol Ther. 2022;35(11). doi:10.1111/dth.15868
- [Background] Mahmoudi H, Daneshpajooh M, Dadkhahfar S, et al. Efficacy and safety of tofacitinib in the treatment of adults with lichen planopilaris: A randomized placebo-controlled trial. Int Immunopharmacol. 2025;162:115129. doi:10.1016/j.intimp.2025.115129
- [Background] Rácz E, Gho C, Moorman PW, Noordhoek Hegt V, Neumann HAM. Treatment of frontal fibrosing alopecia and lichen planopilaris: a systematic review. J Eur Acad Dermatology Venereol. 2013;27(12):1461-1470. doi:10.1111/jdv.12139
- [Background] Husein-ElAhmed H, Husein-ElAhmed S. A Systematic Review and Bayesian Network Meta-Analysis of Medical Therapies for Lichen Planopilaris. Dermatology. 2024;240(1):103-110. doi:10.1159/000534364
- [Background] Valdez-Zertuche JA, Ramírez-Marín HA, Tosti A. Efficacy, safety and tolerability of drugs for alopecia: a comprehensive review. Expert Opin Drug Metab Toxicol. 2025;21(4):347-371. doi:10.1080/17425255.2025.2461483
- [Background] Svigos K, Yin L, Fried L, Lo Sicco K, Shapiro J. A Practical Approach to the Diagnosis and Management of Classic Lichen Planopilaris. Am J Clin Dermatol. 2021;22(5):681-692. doi:10.1007/s40257-021-00630-7